CLINICAL TRIAL: NCT01346475
Title: A Randomized, Cross-Over Study to Evaluate the Suppressive Effect of High-Dose Valacyclovir Versus Once Daily Valacyclovir on Herpes Simplex Virus Type 2 Genital Shedding in Herpes Simplex Virus-2 Seropositive Adults
Brief Title: Randomized Trial to Evaluate Suppressive Effect of High-Dose Valacyclovir Versus Once-Daily Valacyclovir on Persons With HSV-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Christine Johnston, Acting Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30520-D - Phase 2
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- valacyclovir (Active Comparator)
  Interventions: Drug: Valacyclovir
- high dose valacyclovir (Experimental)
  Interventions: Drug: valacyclovir

INTERVENTIONS:
Drug: valacyclovir — 1000 mg orally three times daily for 5 weeks
  Arms: high dose valacyclovir
Drug: Valacyclovir — 500 mg orally once daily for 5 weeks
  Arms: valacyclovir

SUMMARY:
On 13 August 2008, this trial was submitted to ClinicalTrials.gov as modification to NCT00362297. On 28 April 2011, the two records were split for administrative purposes and each trial was given its own unique study record. Please refer to the "History of Changes" on posting NCT00362297 for a detailed summary of the modifications.

The purpose of the research study is to evaluate the effectiveness of high-dose valacyclovir compared to once daily valacyclovir for reduction of asymptomatic HSV-2 genital shedding in persons with genital herpes.

The study will enroll men and women who are 18 years or older, test positive to HSV-2 (by blood test) and have had a first outbreak of HSV-2 within the past 6 months or have had at least 4 genital herpes outbreaks in the past year. Participants must be HIV negative and willing to stop taking suppressive therapy for HSV for the one week wash out period. (Females only: You must not be pregnant or breast-feeding). Both men and women will be asked to use an effective form of birth control.

Involvement in the study will last 11-weeks and you will be asked to visit the clinic every 2-weeks. At each visit, you will be given medication to take daily (either once daily valacyclovir or high dose valacyclovir; you will receive both medications at some point during this study). We will ask you to give a blood sample for liver, kidney and blood count testing at each visit. There will be a total of 8 study visits and each visit will last approximately 30 minutes. We will ask that you complete a daily symptom diary and collected daily home swabs 4-times a day, everyday during the study. Each daily home swab will take less than 3 minutes to perform.

DETAILED DESCRIPTION:
Screening Assessment

Patients will be assessed for their eligibility to enter the study at a screening visit. After signing informed consent they will undergo a medical history and the following information will be recorded in the Case Report Form (CRF):

* Demographic Data: Date of birth, sex, marital status, education and race
* Previous antiviral medication taken
* History of sexually transmitted infections and sexual history.
* Women of childbearing potential will undergo a urine pregnancy test. Serologic samples for HSV-2 and HIV will be obtained. Part of the blood sample will also be used for safety labs.

Start of Study Visit (Day 0) and Day 14, 28, 35, 42, 56, 70, and 77 Follow-Up Visits.

Eligible patients will return to clinic to be given study drug and a patient diary card on which to record concomitant medications, signs and symptoms, and adverse experiences. The investigator will instruct the patient on daily home viral sample collection, taking the study drug, and completing the diary card. The patient will be instructed to return to clinic in 2 weeks, +/- 2 days. Medication compliance will be assessed at each visit using pill counts. Safety labs will be performed on day 14, 28, 35, 56, 70 and 77.

Crossover Study Visit Prior To Washout Period (Day 35-41)

Participants will not be given study drug or placebo during the 7-day washout period. Participants will not be required to obtain swabs during the washout period.

Daily Home Viral Sample Collection

Participants will collect swabs from the genital mucosa four times per day and store the samples in PCR media with preprinted labels. Women will swab the cervicovaginal, vulvar and perianal areas, and men will swab the penile and perianal. Every two weeks, they will return the samples to the Virology Research Clinic when they present for additional study drug and assessment.

Final Study Visit (Day 77)

At the final study visit at Day 77 or for premature discontinuation, the investigator will perform the activities at the regular study visits, with the exception of the dispensation of study drug.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* HSV-2 seropositive by Western Blot;
* not receiving any drugs with known anti-HSV-2 activity for study duration;
* history of primary genital herpes infection within past 6 months OR history of 4 or more HSV recurrences per year during the past year OR 4 or more recurrences per year prior to initiation of suppressive antiviral therapy; or shedding HSV-2 from genital mucosa on >25% of days in shedding session performed at the VRC within the last 2 years.
* able to comply with the study protocol;
* women of child bearing potential who are sexually active with men must be using a medically accepted method of contraception as judged by the investigator;
* women of child-bearing potential must have a negative pregnancy test (urine) at screening visit;
* in general good health, without other serious medical conditions and specifically with normal renal and hepatic function, as determined by the patient's medical history;
* planning to remain resident in the area of the study center for the duration of the study participation;
* HIV seronegative.

Exclusion Criteria:

* hypersensitivity to acyclovir or valacyclovir;
* pregnant women;
* HIV positive or other immunosuppressed state, including chronic steroid use. Intermittent nasal or topical steroids are acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Johnston, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Derived] Johnston C, Saracino M, Kuntz S, Magaret A, Selke S, Huang ML, Schiffer JT, Koelle DM, Corey L, Wald A. Standard-dose and high-dose daily antiviral therapy for short episodes of genital HSV-2 reactivation: three randomised, open-label, cross-over trials. Lancet. 2012 Feb 18;379(9816):641-7. doi: 10.1016/S0140-6736(11)61750-9. Epub 2012 Jan 4. PMID 22225814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from October 2008 to April 2010. Participants recruited at the University of Washington Virology Research Clinic in Seattle, WA.
Groups:
- Standard-dose Valacyclovir First Then High-dose Valacyclovir: Standard-dose valacyclovir (500 mg daily) for 5 weeks followed by 1 week wash-out and then high-dose valacyclovir (1 gram three times daily) for 5 weeks
- High-dose Valacyclovir First Then Standard-dose Valacyclovir: High-dose valacyclovir (1 gram three times daily) for 5 weeks followed by 1 week wash-out and then standard-dose valacyclovir (500 mg daily) for 5 weeks
Period: First Intervention
Arm/Group | Standard-dose Valacyclovir First Then High-dose Valacyclovir | High-dose Valacyclovir First Then Standard-dose Valacyclovir
Started | 22 | 28
Completed | 18 | 25
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3
Period: Second Intervention
Arm/Group | Standard-dose Valacyclovir First Then High-dose Valacyclovir | High-dose Valacyclovir First Then Standard-dose Valacyclovir
Started | 18 | 25
Completed | 18 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | High Dose Valacyclovir | Total
Number analyzed (Participants) | 22 | 28 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (9.5) | 37.7 (12.8) | 40.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 9 | 13 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 18 | 25 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of HSV-2 Total Shedding From the Genital Tract as Measured by PCR, Calculated Using a Per-day Shedding Rate in Participants Treated With High-dose Valacyclovir as Compared to Once-daily Valacyclovir.
Time Frame: 11 weeks
Population: Participants who collected at least one swab on each arm of the cross-over were included in the analysis.
Measure: Number; unit: percentage of swabs with HSV detected
Units Other Than Participants: Swabs
Arm/Group | Standard-dose Valacyclovir (500 mg Daily) | High-dose Valacyclovir (1 gm Three Times Daily)
Number analyzed (Participants) | 43 | 43
Number analyzed (Swabs) | 5008 | 4973
percentage of swabs with HSV detected | 5 | 3
Statistical Analysis 1: Comparison: Standard-dose Valacyclovir (500 mg Daily) vs High-dose Valacyclovir (1 gm Three Times Daily); This study had 80% power to detect a 50% reduction in HSV genital shedding rates for high-dose valacyclovir compared to standard dose valacyclovir; Test type: Superiority or Other; p < 0.001, Incident risk ratio; The model is adjusted for period effects; Incident Risk Ratio = 0.54, 95% CI 2-sided [0.44 to 0.66]

2. Secondary Outcome: Quantity of HSV Detected, Median
Description: Median quantity of HSV detected, among swabs with any HSV detected
Time Frame: 11 weeks
Measure: Median (Inter-Quartile Range); unit: log 10 copies/ml
Units Other Than Participants: swabs
Arm/Group | Standard-dose Valacyclovir (500 mg Daily) | High-dose Valacyclovir (1 gm Three Times Daily)
Number analyzed (Participants) | 43 | 43
Number analyzed (swabs) | 292 | 164
log 10 copies/ml | 3.0 [2.4 to 4.5] | 2.5 [2.3 to 2.7]

3. Secondary Outcome: Number of Genital HSV Shedding Episodes
Description: The number of HSV shedding episodes. A shedding episode is defined as any number of positive swabs preceded and followed by 2 negative swabs.
Time Frame: 11 weeks
Measure: Number; unit: Episodes
Arm/Group | Standard-dose Valacyclovir (500 mg Daily) | High-dose Valacyclovir (1 gm Three Times Daily)
Number analyzed (Participants) | 43 | 43
Episodes | 58 | 65

4. Secondary Outcome: Duration of Genital HSV Shedding Episodes
Description: Median duration of HSV shedding episodes, in hours, among episodes of known duration
Time Frame: 11 weeks
Measure: Median (Inter-Quartile Range); unit: Hours
Units Other Than Participants: Episodes
Arm/Group | Standard-dose Valacyclovir (500 mg Daily) | High-dose Valacyclovir (1 gm Three Times Daily)
Number analyzed (Participants) | 43 | 43
Number analyzed (Episodes) | 42 | 41
Hours | 10 [7 to 42] | 7 [6 to 9]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the 11 week study period.
Description: Adverse event data was collected on 43 participants who completed the trial. In addition, 1 participant who withdrew during the standard dose valacyclovir arm and 1 participant who withdrew during the high dose valacyclovir arm had adverse events, and these data are included in the total number of AEs and participants included.
Arm/Group | Valacyclovir | High Dose Valacyclovir
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 2/44 | 20/44
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=44) | High Dose Valacyclovir (N=44)
Headache (Nervous system disorders) | 0 (0) | 13
Nausea (Gastrointestinal disorders) | 0 (0) | 3
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
This trial was performed at a single site and enrolled healthy, mostly white adults with frequent genital herpes outbreaks. Whether these finding are generalizable to other populations is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review and comment on any proposed publication, and all Study results and data reasonably necessary for a meaningful review of the proposed publication are submitted to the sponsor for a period of at least thirty (30) days prior to submitting the publication to any third party.